CLINICAL TRIAL: NCT00738517
Title: Immunoadsorption With Subsequent Immunoglobulin Substitution for Patients With Heart Failure After Myocardial Infarction
Brief Title: Immunoadsorption and Immunoglobulin Substitution for Heart Failure After Myocardial Infarction
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI left center
Sponsor: University Medicine Greifswald (Other)
Collaborators: Fresenius Medical Care North America (Industry)
Responsible Party: Dr. med. L. R. Herda, Ernst-Moritz-Arndt-Universität
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPG 01/08
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Heart Failure; Coronary Heart Disease
Keywords: heart failure; coronary heart disease; autoantibodies; immunoadsorption; immunoglobulin substitution
MeSH Terms: conditions — Heart Failure; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Immunoadsorption with subsequent immunoglobulin substitution
  Interventions: Device: Immunoadsorption / Immunoglobulin substitution
- 2 (No Intervention)

INTERVENTIONS:
Device: Immunoadsorption / Immunoglobulin substitution — Immunoadsorption with protein-A columns on five consecutive days with subsequent human polyclonal immunoglobulin G substitution after day 5 (0,5g /kg bodyweight)
  Other Names: Immunosorba
  Arms: 1

SUMMARY:
The purpose of this study is to investigate, if immunoadsorption of autoantibodies with subsequent substitution of immunoglobulins is able to improve cardiac function of patients with heart failure after myocardial infarction and presence of cardiac autoantibodies.

DETAILED DESCRIPTION:
Heart failure due to coronary heart disease (CHD) remains one of the most frequent causes of death. Left-ventricular ejection fraction < 30% is associated with a 5-year mortality > 70%. Therefore, new strategies and therapies towards treatment of heart failure are needed.

Heart failure due to left ventricular dysfunction can develop in CHD beyond the area of myocardial infarction. Some of these patients develop myocardial autoantibodies, which have been shown to exert a negative inotropic effect. Their elimination by immunoadsorption has been shown to improve left ventricular function in dilatative cardiomyopathy. Immunoglobulins are substituted to minimize infection risk at a level, which has been shown not to effect cardiac function. This intervention might also ameliorate cardiac function in patients with heart failure due to other origins. This study therefore aims to evaluate the effect of immunoadsorption with subsequent immunoglobulin substitution.

ELIGIBILITY:
Inclusion Criteria:

* heart failure and known coronary heart disease / post myocardial infarction
* completed treatment for coronary heart disease (no known hemodynamically effective stenosis in coronary vessels)
* evidence of scarred myocardial tissue in low-dose stress echocardiography or myocardial scintigraphy or MRI
* evidence of hypo-contractile myocardium in echocardiography or MRI outside of infarction area
* at least 3 months without acute coronary syndrome or coronary intervention
* left-ventricular ejection fraction by echocardiography < 45%
* detection of at least one myocardial autoantibody (e.g. anti-ß1-receptor, anti-TnI, anti-KchIP2) in serum
* dyspnea on exertion equivalent to NYHA II - NYHA IV
* written informed consent of the patient

Exclusion Criteria:

* heart failure due to other cardiac disease (e.g. dilatative cardiomyopathy without evidence of CHD, primary valve defects > II°, toxic cardiomyopathy)
* active infection
* pregnancy
* malign tumor disease
* other secondary disease with life expectancy < 1 year
* refusal by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
left-ventricular ejection fraction as measured by echocardiography | 6 months

SECONDARY OUTCOMES:
cardiac index | 6 months
systemic vascular resistance | 6 months
pulmonary vascular resistance | 6 months
n-terminal pro-BNP concentration (serum) | 6 months
peak oxygen uptake (spiroergometric) | 6 months
dyspnoea symptoms / NYHA classification | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephan B Felix, MD, Study Chair — University Medicine Greifswald; Lars R Herda, MD, Study Director — University Medicine Greifswald; Astrid Hummel, MD, Principal Investigator — University Medicine Greifswald; Marcus Doerr, MD, Principal Investigator — University Medicine Greifswald; Daniel Beug, MD, Principal Investigator — University Medicine Greifswald
Locations (1):
- Ernst-Moritz-Arndt-Universität, Greifswald, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Background] Jahns R, Boivin V, Siegmund C, Inselmann G, Lohse MJ, Boege F. Autoantibodies activating human beta1-adrenergic receptors are associated with reduced cardiac function in chronic heart failure. Circulation. 1999 Feb 9;99(5):649-54. doi: 10.1161/01.cir.99.5.649. PMID 9950662
- [Background] Okazaki T, Tanaka Y, Nishio R, Mitsuiye T, Mizoguchi A, Wang J, Ishida M, Hiai H, Matsumori A, Minato N, Honjo T. Autoantibodies against cardiac troponin I are responsible for dilated cardiomyopathy in PD-1-deficient mice. Nat Med. 2003 Dec;9(12):1477-83. doi: 10.1038/nm955. Epub 2003 Nov 2. PMID 14595408
- [Background] Dorffel WV, Felix SB, Wallukat G, Brehme S, Bestvater K, Hofmann T, Kleber FX, Baumann G, Reinke P. Short-term hemodynamic effects of immunoadsorption in dilated cardiomyopathy. Circulation. 1997 Apr 15;95(8):1994-7. doi: 10.1161/01.cir.95.8.1994. PMID 9133505
- [Background] Felix SB, Staudt A, Dorffel WV, Stangl V, Merkel K, Pohl M, Docke WD, Morgera S, Neumayer HH, Wernecke KD, Wallukat G, Stangl K, Baumann G. Hemodynamic effects of immunoadsorption and subsequent immunoglobulin substitution in dilated cardiomyopathy: three-month results from a randomized study. J Am Coll Cardiol. 2000 May;35(6):1590-8. doi: 10.1016/s0735-1097(00)00568-4. PMID 10807465
- [Background] Staudt A, Schaper F, Stangl V, Plagemann A, Bohm M, Merkel K, Wallukat G, Wernecke KD, Stangl K, Baumann G, Felix SB. Immunohistological changes in dilated cardiomyopathy induced by immunoadsorption therapy and subsequent immunoglobulin substitution. Circulation. 2001 Jun 5;103(22):2681-6. doi: 10.1161/01.cir.103.22.2681. PMID 11390337